CLINICAL TRIAL: NCT06139848
Title: Comparison of Posterior -Anterior Spinal Mobilization and Prone Press up on Pain ,Range of Motion and Disability in Patients With Non Specific Low Back Pain.
Brief Title: Comparison of Posterior-anterior Spinal Mobilization and Prone Press up in Patients With Non Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCRAHS-ISB-REC/MS-PT-01609
Record Dates: First submitted 2023-09-15; First posted 2023-11-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Non-specific Low Back Pain
Keywords: Non specific low back pain; Range of motion; Disability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maitland, Mackenzie Techniques and Conventional Treatment (Experimental): posterior-anterior spinal mobilization and prone press up along with conventional treatment as Heating pad for 10 minutes Bridging exercises (10 rep, 3 sets) Paraspinal muscle stretch
  Interventions: Other: Posterior-anterior spinal mobilization, prone press up Techniques
- Maitland Mobilization Techniques and Conventional Treatment (Active Comparator): Posterior-anterior spinal mobilization along with conventional treatment as Heating pad for 10 minutes Bridging exercises (10 rep, 3 sets) Paraspinal muscle stretch
  Interventions: Other: Traditional Physical Therapy
- Meckinzie Techniques and Conventional Treatment (Active Comparator): Prone press up technique will be given along with conventional treatment as:
  Heating pad for 10 minutes Bridging exercises (10 rep, 3 sets) Paraspinal muscle stretch
  Interventions: Other: Traditional Physical Therapy; Other: Posterior-anterior spinal mobilization, prone press up Techniques

INTERVENTIONS:
Other: Traditional Physical Therapy — Conventional therapy include heating therapy for 10 mints, Bridging exercises (10 rep, 3 sets), Paraspinal muscle stretch.
  Other Names: Conventional Therapy
  Arms: Maitland Mobilization Techniques and Conventional Treatment; Meckinzie Techniques and Conventional Treatment
Other: Posterior-anterior spinal mobilization, prone press up Techniques — Posterior-anterior spinal mobilization and prone press- ups techniques. Posterior- Anterior glides and prone press up along with conventional therapy. PA Mobilization on lumber spine, grade I if patient feel no pain the therapist will proceed to grade III-IV. 3 sets for 40 seconds. Total time 10 mints.
  Prone press-ups will be performed actively by the patients without no reproduction of pain with lumber extension in standing. In prone press-up the patient pelvis stabilized in prone position and asked for active extension. End range time 5 seconds. Total 10 repetitions.
  Arms: Maitland, Mackenzie Techniques and Conventional Treatment; Meckinzie Techniques and Conventional Treatment

SUMMARY:
No previous literature found on the comparison of posterior-anterior spinal mobilization and prone press-up on pain, range of motion and disability in patients with non-specific low back pain. This study will approach the results of posterior- anterior spinal mobilization and prone press-up on pain, range of motion and disability in patients with non-specific low back pain. In previous researches the patients were not properly followed to see pre session, immediate after the session and after twenty- four hours effects of both interventions Posterior- anterior mobilization and Press-ups. Secondly, they have not taken the control group in their studies. In current study two techniques along with conventional treatment will be compared in three different groups to see their individual effects and combine effect of Maitland and Mackenzie technique

DETAILED DESCRIPTION:
Non-specific low back pain refers to pain without any specific cause. The term "non- specific low back pain" refers to a condition where the cause of the symptoms cannot be identified with certainty, indicating that the underlying pathology is currently unknown and difficult to diagnose reliably. This pain is known for the main leading cause to effect activities of daily life, absenteeism and health care. Non-specific low back pain is a widely known serious condition in the worldwide . this was a randomized control trial and patients were randomly selected according to inclusion criteria and divided into A and B and C groups. The base line demographic, clinical and disability data was collected through structured questionnaire. Group A received both posterior-anterior mobilization on L4 and L5 level and Prone press- ups technique along with a conventional therapy whether group B had received only posterior-anterior spinal mobilization along with the conventional therapy. While group C received prone press-ups technique along with conventional treatment. Patient outcomes were measured at baseline, immediate after the session and 24 hours after the session outcomes measures (NPRS, GONIOMETER, ODI).

ELIGIBILITY:
Inclusion Criteria:

* Non-specific low back pain of duration <3 months
* Both male and female Age 22-40
* Increased localized pain with lumber extension during standing
* NPRS < 6

Exclusion Criteria:

* Spinal Surgery
* Subject who administered epidural injections
* Psychological low back pain
* History of injury from past 3 months
* Neurological deficit
* Hyper-mobility
* Subjects with mental disorder

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
NPRS (Numeric pain rating scale) | Baseline, after treatment and after 24 hours of session
  NPRS (Numeric pain rating scale) is a scale used to check whether the pain is mild, moderate and severe.
Inclinometer | Baseline, after treatment and after 24 hours of session
  Inclinometer device is used to measure range of motion of the lower back
Oswestory Disability Index | Baseline, after treatment and after 24 hours of session
  Oswestory Disability Index is a measuring tool to collect data from patients. 0-4 shows no disability, 5-14 mild disability, 15-24 moderate disability, 25-34 severe disability, 35-50 reveals completely disabled. it helps to provide data about patient's low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ishtiaq, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Khyber Teaching Hospital Peshawar, Peshawar, Khyber Pakhtun Khwa, Pakistan

IPD SHARING:
Plan to Share IPD: No